CLINICAL TRIAL: NCT06331078
Title: Comparison of the Effects of Square Step Exercises and Aerobic Exercise on Cognitive Functions and Physical Fitness in Healthy Young Adults
Brief Title: Square Step Exercises in Healthy Young Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Ezgi Eryildiz, MSc, PT, Research Assistant, Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 29.02.2024/45
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-03

CONDITIONS: Exercise; Square Step Exercises; Aerobic Exercise; Cognitive Function; Physical Fitness
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Square Stepping Exercise Group (Experimental): The experimental group will have Square Stepping Exercise training twice a week for 4 weeks. Each session will start with a 15-minute warm-up, followed by a 40-minute Square Stepping Exercise workout and ending with a 15-minute cool-down. The Square Stepping Exercise part will start with the Elementary 2 level, which has 30 different patterns. Participants will start with the first pattern at this level. If they can complete it without mistakes within 15 seconds, they'll move on to the next pattern. If not, they'll repeat the pattern until they get it right within the time limit. Each session will have four participants, with two participants working on each of the two mats, which are divided into 40 squares and measure 100cm by 250 cm.
  Interventions: Other: Square Stepping Exercise training
- Aerobic Exercise Group (Active Comparator): Individuals in the aerobic control cohort will partake in a 40-minute treadmill walking session, maintaining their heart rate at 60% of their individual heart rate reserve as calculated using the Karvonen formula. Before and after the aerobic exercise, a 5-minute warm-up session incorporating stretching and calisthenics, as well as a 5-minute cool-down session, will be conducted.
  Interventions: Other: Aerobic Exercise Training

INTERVENTIONS:
Other: Square Stepping Exercise training — The experimental group will have Square Stepping Exercise training.
  Arms: Square Stepping Exercise Group
Other: Aerobic Exercise Training — Individuals in the aerobic control cohort will partake in a treadmill walking session.
  Arms: Aerobic Exercise Group

SUMMARY:
This study aims to compare the effectiveness of Square Stepping Exercise and aerobic exercise on cognitive function and physical fitness in young adults. Participants aged 18-30 with low physical activity levels will be randomly assigned to either the Square Stepping Exercise Group or Aerobic Exercise Group. Both interventions will be supervised by a physiotherapist, performed twice a week for 40 minutes over 4 weeks. Cognitive function will be assessed using various tests, including attention, short-term memory, and executive function evaluations. Physical fitness will be evaluated through jump tests and balance assessments. Blinded assessors will conduct evaluations at baseline and post-intervention in both groups to determine the impact of square stepping exercise and aerobic exercise on cognitive and physical health in young adults.

ELIGIBILITY:
Inclusion Criteria:

* International Physical Activity Questionnaire score <600 Metabolic Equivalents (METs),
* No neurological or orthopedic problems affecting gait, balance and lower extremities
* No vision or hearing problems, and no history of musculoskeletal surgery.

Exclusion Criteria:

* Participants who have pain due to a musculoskeletal problem
* Participants who are continuing another routine exercise program

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Schulte Grid Test | Baseline and after the interventions (4th week)
  Schulte Grid Test will be used to evaluate the attention level of the participants. The task involves participants locating and selecting numbers in sequential order within a table filled with random numbers ranging from 1 to 64. Participants are required to find and click the correct numbers in ascending order, with completion time serving as the primary metric for assessment. Once a participant selects the correct number "1," the corresponding box will illuminate in green, prompting the participant to locate and select "2," and so forth until reaching "64." The test concludes upon successfully clicking the last number in the sequence. Schulte grid test will be conducted on a 15.6-inch laptop screen. A shorter reaction and completion time for the test will show good attention.
Stroop Test | Baseline and after the interventions (4th week)
  This test will be used to evaluate executive functions, particularly selective attention and cognitive flexibility. In this assessment, participants are tasked with identifying the colors of rectangles, reading color names, and stating the color of color names printed in differing hues. Subsequently, error rates and spontaneous corrections are meticulously recorded and assessed. A shorter completion time and fewer number of errors for the test will show good executive functions.
Verbal Fluency Test | Baseline and after the interventions (4th week)
  1. Letter Fluency Test: Participants are instructed to count words beginning with the letters K, A, S, and non-numerical characters within one minute, while a voice recording is made. Words not starting with the specified letters and repeated words are tallied as errors/points. It is scored on the number of words derived. Repetition of the same word is considered as perseveration
  2. Category Fluency Test: Participants are prompted to enumerate names of animals, fruits, and objects purchasable from the market within one minute, with a voice recording taken. Words falling outside the designated categories and repetitions are logged as error count/score. Total score based on the number of groups formed by the individual in one minute points are awarded. The more groups the individual has made, the more points individual gets.
  In this study, these tests will be utilized to assess information processing speed and attention as part of executive functions.
Digit Span Test | Baseline and after the interventions (4th week)
  The test consists of two parts. Part One is Digits Forward and Part Two is Digits Backward. In both tests administered separately, random numbers are read to the participants at one-second intervals. The norm value of the Digits Forward is 7, while the norm value of the Digits Backward is 5; results below these values indicate impaired attention.
Vertical jump test | Baseline and after the interventions (4th week)
  This test will be used for physical fitness assessment. During the assessment, the participant positions themselves adjacent to a wall. Using one arm, they extend upwards without bending, making contact with a wall marked in centimeters (cm). This measurement is then recorded. Following this, the participant is directed to perform a maximal force jump, aiming to touch the highest point achievable. This process is repeated thrice, with a 60-second rest interval between each jump. The highest value attained among the three jumps is documented in centimeters.
Horizontal jump test | Baseline and after the interventions (4th week)
  In the assessment of horizontal jump, a key component of physical fitness, the standing long jump technique will be utilized. A designated starting line will be marked, with a ruler spanning 3 meters in length fixed at 1-centimeter intervals from the starting point. Participants will assume the starting position, ensuring their feet are not touching the line and are fully grounded, then execute a forward jump using both legs. The distance from the starting line to the point where the participant's feet last touch the ground will be measured. Each participant will perform three jumps, and the best distance achieved will be recorded as the final measurement.
Y Balance Test | Baseline and after the interventions (4th week)
  Dynamic balance, an essential component of physical fitness crucial for executing functional tasks and occupational activities, will be evaluated using the Y balance test. This test involves reaching as far forward as possible along anterior, posterolateral, and posteromedial directional lines placed on the ground while maintaining balance on one foot. Participants will be instructed to reach as far as they can in each direction with their raised foot while keeping their hands on their hips. The maximum reach distances achieved in the anterior, posteromedial, and posterolateral directions will be marked and recorded as three valid measurements for each direction. The key outcome measures of interest will include the reach distances in the three directions as well as the composite score derived from the test.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No